CLINICAL TRIAL: NCT05444296
Title: Superficial Dry Needling of the Trigeminal Nerve Innervation Sensory Field for Cervicogenic Headache: a Randomized Clinical Trial
Brief Title: Superficial Dry Needling for Cervicogenic Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Youngstown State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-186
Record Dates: First submitted 2022-06-27; First posted 2022-07-05 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Intervention Model Description: Single blinded, randomized, active control
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blind to the type of intervention the participant receives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): Experimental group
  Interventions: Other: Superficial Dry Needling; Other: Non-thrust Mobilizations only
- Upper Cervical Mobilizations (Active Comparator): Active control
  Interventions: Other: Non-thrust Mobilizations only

INTERVENTIONS:
Other: Superficial Dry Needling — 1/2" needles will placed into defined innervation fields of the trigeminal nerve and rotated. Total time will be 5-7 minutes.
  Other Names: Non-thrust mobilizations
  Arms: Dry Needling
Other: Non-thrust Mobilizations only — Non-thrust mobilizations to be applied to the most symptomatic level of the upper cervical spine as determined by a treating physical therapist. The mobilization technique will be applied for 3 bouts of 30 seconds.

SUMMARY:
It is unknown if applying superficial dry needling to the trigeminal innervation field improves pain and disability for patients with cervicogenic headaches. The aim of this study is to determine if superficial dry needling of the trigeminal innervation field improves pain, neck mobility, and disability in patients with cervicogenic headaches. It will also be examined if psychosocial factors such as stress, anxiety, depression and self efficacy influence improvements in pain, range of motion and neck disability.

DETAILED DESCRIPTION:
Cervicogenic headache (CGH), is defined by the International Classification of Headache Disorders (ICHD) as a "headache caused by a disorder of the cervical spine and its component bony, disc, and/or soft tissue elements, usually but not invariably accompanied by neck pain. Prevalence of CGH in the general population is between .4-20%. Although the primary source of pain is generated from the upper cervical spinal levels, there is also neuro-anatomical basis of CGH involving the trigeminal nerve.

Dry needling (DN) is a widely used intervention performed by physical therapists for a wide range of musculoskeletal and neurological conditions. Dry needling has been shown to be beneficial for CGH but DN has only been investigated using trigger point DN to cervical musculature. Superficial DN also reduces pain associated to orthopedic spinal conditions and may be associated with a lower risk of post-treatment soreness.

Non-thrust mobilizations of the cervical spine are an accepted treatment known to reduce pain and disability associated with CGH. Their use has also been recommended in clinical practice guidelines.

This study aims to look investigate whether superficial dry needling targeting the trigeminal innervation sensory field will reduce pain and impairments known to exist in patients with CGH compared to mobilizations of the cervical spine. Mobilizations of the cervical spine are another common treatment that physical therapists employ to treat cervicogenic headaches.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Symptoms: (1)Unilateral pain starting in the neck and radiating to the frontotemporal region or posterior fossa, (2) pain aggravated by neck movement, (3) restricted cervical range of motion, (4) non-throbbing and non-lancinatingnpain, 5) dysfunction/headache pain in at least one of the joints of the upper cervical spine(C0-C4), and (6) headache frequency of at least 1 per week over a period greater than 3 months.

Exclusion Criteria:

* Headache or neck pain <2/10
* Contraindications to the interventions
* Whiplash associated disorder within 6 weeks
* Pending litigation for neck pain and/or headache.
* Unwilling to cease other care through duration of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2022-07-05 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Headache or neck pain intensity on a Numeric pain rating scale (0-10) | <1 hour
  0-10 scale pain intensity, 0 is no pain, 10 is severe pain, the lower the score the better

SECONDARY OUTCOMES:
Flexion Rotation Test in degrees of measurement | <1 hour
  Flexion-rotation test for CGH will be measured to determine any change in measure for c1-c2 mobility.
Active Range of Motion of the Cervical Spine in degrees of measurement | <1 hour
  Active range of motion will be measured in the most painful and or limited plane of movement.
Patient Health Questionnaire - 9 (PHQ-9) | <1 hour
  Patient Health Questionnaire-9 is used to assess the severity of depression an individual may have. It is scored from 1-27. The lower the score, the lower the severity of depression an individual has.
Short Form 36 (SF-36) | <1 hour
  Short Form-36 is used to assess quality of life. Each section of the Short Form 36 is scored with weight scores from 0-100. There is specific coding per section to assess different aspects of quality of life, for example physical functioning, emotional wellbeing. 100 in each section indicates a person is functioning at the highest level possible.
Generalized Anxiety Disorder 7 (GAD-7) | <1 hour
  Generalized Anxiety Disorder-7 is used to assess the severity of anxiety an individual may have. The Generalized Anxiety Disorder 7 is scored from 0-21. A lower score indicates less severity of anxiety.
Neck Disability Index (NDI) | <1 hour
  Neck Disability Index is used to assess how much an individual's neck pain affects daily life. The Neck Disability Index is scored from 0-50 and transformed into a percentage. This indicates the amount of disability someone has. The lower the score, the less disability is caused by neck pain.
Headache Self Efficacy Scale (HSES) | <1 hour
  Headache Self Efficacy Scale is used to assess an individual's belief they can do things to prevent headaches. Higher scores indicate higher self efficacy. The items have scoring from 1-7 with 1 being strongly disagree and 7 being strongly agree. Some items are reverse scored. The scores can range from 79-121.
Injection Phobia Scale (IPS) | <1 hour
  The Injection Phobia Scale assesses a person's fear or anxiety toward injections. It is scored 0-32 with the higher score indicating more severity of a phobia of injections.
Severity Measure for Specific Phobia-Adult (SMSP-A) | <1 hour
  The Severity Measure for Specific Phobia-Adult assesses symptoms a person feels in response to injections and/or needles. It is scored 0-40 with higher scores indicating more severity of phobia of needles.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Learman, PhD, Study Director — Director of the PhD in Health Sciences
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vazquez-Justes D, Yarzabal-Rodriguez R, Domenech-Garcia V, Herrero P, Bellosta-Lopez P. Effectiveness of dry needling for headache: A systematic review. Neurologia (Engl Ed). 2020 Jan 13:S0213-4853(19)30144-6. doi: 10.1016/j.nrl.2019.09.010. Online ahead of print. English, Spanish. PMID 31948718
- [Background] Gildir S, Tuzun EH, Eroglu G, Eker L. A randomized trial of trigger point dry needling versus sham needling for chronic tension-type headache. Medicine (Baltimore). 2019 Feb;98(8):e14520. doi: 10.1097/MD.0000000000014520. PMID 30813155
- [Background] France S, Bown J, Nowosilskyj M, Mott M, Rand S, Walters J. Evidence for the use of dry needling and physiotherapy in the management of cervicogenic or tension-type headache: a systematic review. Cephalalgia. 2014 Oct;34(12):994-1003. doi: 10.1177/0333102414523847. Epub 2014 Mar 12. PMID 24623124